CLINICAL TRIAL: NCT02675530
Title: Parallel Effects of Ketamine and Schizophrenia on Neurocognitive Function
Brief Title: Parallel Effects of Schizophrenia and N-methyl-D-aspartate (NMDA) Antagonism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 0612002073
Record Dates: First submitted 2012-05-17; First posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Schizophrenia
Keywords: NMDA; glutamate; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy control (Experimental): Healthy controls will receive electrophysiological assessments before and after NMDA antagonist administration.
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: ketamine — For healthy volunteer arm of study, NMDA antagonist ketamine will be administered. 0.23 mg/kg over 1 minute, followed by 0.58 mg/kg/hour for 30 minutes, followed by 0.29 mg/kg/hour for 50 minutes.
  No drug administration for patients with schizophrenia

SUMMARY:
This study investigates the common features of electrophysiological measures in schizophrenia and effects of NMDA antagonist ketamine in healthy volunteers.

ELIGIBILITY:
Subjects for the Ketamine experiment(Healthy control experiment):

Inclusion Criteria:

1. Male or female
2. 21-45 years old
3. Deemed healthy by the Structured Clinical Interview for DSM-NP (SCID-NP) and collateral information. Subjects will need to provide the name of a person, preferably a family member, whom the research team can contact to corroborate information.

Exclusion Criteria:

1. Lifetime diagnosis of DSM-IV substance dependence (except caffeine and nicotine).
2. Substance abuse, as per clinical judgment, in the past 1 year.
3. Current or past DSM-IV Axis-I diagnosis.
4. A history of significant medical/neurological disease such as cardiac, thyroid, renal, hepatic or neurological. Unstable medical condition based on EKG, vital signs, physical examination and laboratory work-up.
5. A hearing deficit greater than 30 dB in both ears detected using a Welch-Allyn audioscope (500, 1000, 2000 and 4000 Hz threshold will be evaluated) at screening.
6. Major current or recent (<6 weeks) stressors.
7. History of counseling, except if counseling was for a life circumstance disorder (e.g., bereavement, divorce) or in the opinion of the investigator, is not clinically significant.
8. Lifetime history of treatment with any psychotropic medications for > 1 month duration suggestive of psychiatric illness.
9. Current or past Axis I diagnosis of schizophrenia or bipolar disorder in first-degree relatives.
10. Any medication that could interfere with either the safety of the study and/or the outcome measures.
11. Use of any illicit substances in the 4 weeks prior to beginning study participation.
12. Any history indicating learning disability, mental retardation, or attention deficit disorder.
13. History of head injury with loss of consciousness greater than fifteen minutes.
14. Any other condition or medication, which in the opinion of the investigator would preclude participation in the study.
15. Non-English speaking.
16. Known sensitivity to ketamine.

Subjects for the Schizophrenia experiment:

Inclusion Criteria for control subjects:

1. Male or female
2. 21-45 years old
3. No past or present Axis I diagnosis, as determined by the SCID-NP

Exclusion Criteria for control subjects:

1. Lifetime diagnosis of DSM-IV substance dependence (except caffeine and nicotine).
2. Substance abuse, as per clinical judgment, in the past 1 year
3. A history of significant medical/neurological disease such as cardiac, thyroid, renal, hepatic or neurological.
4. A hearing deficit greater than 30dB in both ears detected using a Welch-Allyn audioscope (500, 1000, 2000 and 4000 Hz threshold will be evaluated) at screening.
5. Axis I diagnosis of schizophrenia or bipolar disorder in first-degree relatives.
6. History of head injury with loss of consciousness greater than fifteen minutes
7. Any other condition or medication, which in the opinion of the investigator would preclude participation in the study.
8. Non-English speaking.

Inclusion Criteria for patients:

1. Male or female
2. 21-45 years old
3. Diagnosed with DSM-IV schizophrenia based on a SCID-IP interview for patients.
4. Stable dose of antipsychotic medications for at least 2 weeks prior to beginning study participation.
5. Score either in the 1-3 (high functioning) range or in the 5-7 (low functioning) range of the Global Functioning Scale from the MSIF based on a screening interview.

Exclusion Criteria:

1. Lifetime diagnosis of DSM-IV substance dependence (except caffeine and nicotine).
2. Substance abuse, as per clinical judgment, in the past 1 year
3. A history of significant medical/neurological disease such as cardiac, thyroid, renal, hepatic or neurological.
4. A hearing deficit greater than 30dB in both ears detected using a Welch-Allyn audioscope (500, 1000, 2000 and 4000 Hz threshold will be evaluated) at screening.
5. History of head injury with loss of consciousness greater than fifteen minutes.
6. Any other condition or medication, which in the opinion of the investigator would preclude participation in the study.
7. Non-English speaking.

   -

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2007-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
P300, an ERP measure | Baseline and repeat assessment following ketamine

SECONDARY OUTCOMES:
(Mismatch Negativity) MMN | Baseline and repeat assessment

CONTACTS AND LOCATIONS:
Overall Officials: Handan Gunduz-Bruce, M.D., Principal Investigator — Yale Medical School
Locations (1):
- VHA CT, West Haven, Connecticut, United States